CLINICAL TRIAL: NCT02454946
Title: The Relation Between ABO Blood Types and Erectile Dysfunction
Brief Title: Blood Types and Erectile Dysfunction
Status: Completed | Type: Observational
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Erdal Benli, assistant professor, Ordu University
Other Study IDs: ERDL-27
Record Dates: First submitted 2015-05-13; First posted 2015-05-27 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Erectile Dysfunction
Keywords: Blood Group Antigens; erectile dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The researchers aimed to investigate the relationship between ABO blood types and erectile dysfunction.

DETAILED DESCRIPTION:
This retrospective study is done in Ordu university Hospital among patients who administered to urology polyclinic between April 2013 and April 2014. Sexually active 102 patients whose blood types were known were included in this study. While 56 patients had sexual intercourse problems 46 had not and this group was taken as a control group. Individuals who had a sexual partner and whose sexual intercourse were continuing unproblematic ally were accepted as normal. Individuals who had not have sexual intercourse though having a sexual partner or unable to maintain the intercourse were accepted to have sexual dysfunction. Patients' sexual function was evaluated via the İEFF-5 questioning form. In the same session the patients' blood types were also recorded and their İEFF-5 (Erectile Function International Evaluation Form) symptom scores were compared with their blood types.

ELIGIBILITY:
Inclusion Criteria:

* Male, person who have sexual intercourse

Exclusion Criteria:

* Female, who have no sexual intercourse

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Administered to urology polyclinic between April 2013 and April 2014. Sexually active 102 patients whose blood types were known were included in this study.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The relationship between erectile dysfunction and blood group antigens | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin kaya, doctor, Principal Investigator — researcher

REFERENCES:
- [Result] Kaya A, Tanboga IH, Kurt M, Isik T, Kaya Y, Gunaydin ZY, Aksakal E. Relation of ABO blood groups to coronary lesion complexity in patients with stable coronary artery disease. Anadolu Kardiyol Derg. 2014 Feb;14(1):55-60. doi: 10.5152/akd.2013.4728. Epub 2013 Dec 9. PMID 24342931